CLINICAL TRIAL: NCT01893359
Title: A Multi-Center, Randomized, Controlled Evaluation of the Safety and Efficacy of LASIK With Cross-linking Performed With the KXL System and Photrexa ZD™ (Riboflavin Ophthalmic Solution) Compared to LASIK Alone for Hyperopia and Hyperopic Astigmatism
Brief Title: Safety and Efficacy of Corneal Collagen Cross-linking Following LASIK for Treatment of Hyperopia and Hyperopic Astigmatism
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KXL-004
Record Dates: First submitted 2013-06-28; First posted 2013-07-09 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Hyperopia; Hyperopic Astigmatism
Keywords: hyperopia; hyperopic astigmatism; cross-linking
MeSH Terms: conditions — Hyperopia; Astigmatism | interventions — Dextrans; Keratomileusis, Laser In Situ

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LASIK followed by Cross-linking (Continuous Wave) (Experimental): Following LASIK, the corneal bed will be thoroughly coated with five drops of riboflavin ophthalmic solution, rinsed with saline solution, and the corneal flap repositioned. The eye will then be irradiated at 30 mW/cm2 for 2 minutes continuous UVA.
  Interventions: Drug: riboflavin ophthalmic solution, 0% dextran; Device: UVA Irradiation (30 mW/cm2 for 2 minutes continuous UVA); Procedure: Laser-assisted in situ keratomileusis
- LASIK followed by Cross-linking (Pulsed) (Experimental): Following LASIK, the corneal bed will be thoroughly coated with five drops of riboflavin ophthalmic solution, rinsed with saline solution, and the corneal flap repositioned. The eye will then be irradiated at 30 mW/cm2 for 3 minutes pulsed UVA with an on/off cycle of 2 seconds UVA on/1 second UVA off.
  Interventions: Drug: riboflavin ophthalmic solution, 0% dextran; Device: UVA Irradiation (30 mW/cm2 for 3 minutes pulsed UVA with an on/off cycle of 2 seconds UVA on/1 second UVA off); Procedure: Laser-assisted in situ keratomileusis
- LASIK Only (Placebo Comparator): Eyes assigned to this arm will receive standard LASIK with no cross-linking.
  Interventions: Procedure: Laser-assisted in situ keratomileusis

INTERVENTIONS:
Drug: riboflavin ophthalmic solution, 0% dextran
  Other Names: Photrexa ZD
  Arms: LASIK followed by Cross-linking (Continuous Wave); LASIK followed by Cross-linking (Pulsed)
Device: UVA Irradiation (30 mW/cm2 for 2 minutes continuous UVA)
  Other Names: KXL System
  Arms: LASIK followed by Cross-linking (Continuous Wave)
Device: UVA Irradiation (30 mW/cm2 for 3 minutes pulsed UVA with an on/off cycle of 2 seconds UVA on/1 second UVA off)
  Other Names: KXL System
  Arms: LASIK followed by Cross-linking (Pulsed)
Procedure: Laser-assisted in situ keratomileusis
  Other Names: LASIK

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy, with regards to regression of refractive outcome, as measured by manifest refraction spherical equivalent (MRSE), of two treatment regimens for hyperopic and hyperopic astigmatic subjects: LASIK followed by cross-linking performed with the KXL System and Photrexa ZD™ (Riboflavin Ophthalmic Solution), as compared to LASIK alone.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be at least 18 years of age, male or female, of any race;
* 2. Provide written informed consent and sign a HIPAA form;
* 3. Willingness and ability to follow all instructions and comply with the schedule for study visits;
* 4. Undergoing bilateral LASIK for the correction of hyperopia or hyperopic astigmatism;
* 5. Intended treatment > +2.0 diopters (D) to < +6.0 D of MRSE hyperopia or hyperopia with astigmatism, with up to +6.0 D of spherical component and up to 5.0 D of astigmatic component (all refractions measured at the spectacle plane);
* 6. Bilateral physiologic hyperopia;
* 7. For females capable of becoming pregnant, agree to have urine pregnancy testing performed at visit 2 prior to treatment; must not be lactating, and must agree to use a medically acceptable form of birth control for at least one week prior to the visit 2 and continue to use the method for one month following the treatment. Acceptable forms for birth control are spermicide with barrier, oral contraceptive, injectable or implantable method of contraception, transdermal contraceptive, intrauterine device, or surgical sterilization of partner. For non-sexually active females, abstinence will be considered an acceptable form of birth control. Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (e.g. hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
* 8. Best spectacle corrected visual acuity (BSCVA) of 70 letters or more on ETDRS chart;
* 9. Difficulty maintaining uncorrected visual acuity (UCVA) of at least 70 letters on ETDRS chart as evidenced by need for constant contact lens or spectacle wear;
* 10. Less than 0.75 D spherical equivalent difference between cycloplegic and manifest refractions;
* 11. Stable refraction (a difference of 0.50 D or less in MRSE) for the last 12 months, objectively documented (by previous clinical records, prescriptions, etc.), exclusive of changes determined by the investigator to be due to unmasking latent hyperopia;
* 12. Normal corneal topography, as judged by the investigator;
* 13. Removal of contact lenses for the required period of time prior to the screening refraction:

  1. Soft - 3 Days
  2. Soft Toric - 2 Weeks
  3. Rigid gas permeable - 2 Weeks
* 14. Contact Lens Wearers Only: Must demonstrate a stable refraction (a difference of 0.50 D or less) as determined by MRSE on two consecutive exam dates performed at least 7 days apart. A contact lens wearer is defined as someone who has worn contact lenses in either eye in the last 30 days.

Exclusion Criteria:

* 1. Contraindications, sensitivity or known allergy to the use of the test article(s) or their components;
* 2. If female, be pregnant, nursing or planning a pregnancy or have a positive urine pregnancy test at Visit 2 prior to treatment or during the course of the study;
* 3. Eyes which are aphakic;
* 4. Eyes which are pseudophakic and do not have a UV blocking lens implanted;
* 5. Acute or chronic disease or illness that would increase the operative risk or confound the outcomes of the study (e.g., dry eyes, immuno- compromised, connective tissue disease, clinically significant atopic disease, diabetes, etc.);
* 6. Systemic medications that may confound the outcome of the study or increase the risk to the subject, including but not limited to steroids, antimetabolites, etc.;
* 7. Ocular condition that may predispose the subject to future complications, for example:

  1. History or evidence of active or inactive corneal disease (e.g., herpes simplex keratitis, herpes zoster keratitis, recurrent corneal erosion syndrome, corneal dystrophy, etc.);
  2. Evidence of retinal vascular disease;
  3. Keratoconus or keratoconus suspect;
  4. Glaucoma or glaucoma suspect by exam findings and/or family history;
* 8. Previous intraocular or corneal surgery including prior refractive surgery that might confound the outcome of the study or increase the risk to the subject;
* 9. An increased risk for developing strabismus post-treatment;
* 10. Subjects with nystagmus or any other condition that would prevent a steady gaze during treatment or other diagnostic tests;
* 11. Taking supplements containing Vitamin C (ascorbic acid) within 1 week of the cross-linking treatment;
* 12. Corneal thickness <470 microns as measured by Pentacam;
* 13. The Investigator may exclude or discontinue any subject for any sound medical reason;
* 14. The subject should not have participated in any investigational drug or device study within 30 days of screening or be concurrently enrolled in another investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Gordon -Weiss-Schanzlin Vision Institute, San Diego, California
  - Ophthalmic Consultants of Boston, Waltham, Massachusetts
  - Hersh Vision Group, Teaneck, New Jersey
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - See Clearly Vision, McLean, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- LASIK Followed by Cross-linking (Continuous Wave): Following LASIK, the corneal bed will be thoroughly coated with five drops of riboflavin ophthalmic solution, rinsed with saline solution, and the corneal flap repositioned. The eye will then be irradiated at 30 mW/cm2 for 2 minutes continuous UVA.
  riboflavin ophthalmic solution, 0% dextran
  UVA Irradiation (30 mW/cm2 for 2 minutes continuous UVA)
  Laser-assisted in situ keratomileusis
- LASIK Followed by Cross-linking (Pulsed): Following LASIK, the corneal bed will be thoroughly coated with five drops of riboflavin ophthalmic solution, rinsed with saline solution, and the corneal flap repositioned. The eye will then be irradiated at 30 mW/cm2 for 3 minutes pulsed UVA with an on/off cycle of 2 seconds UVA on/1 second UVA off.
  riboflavin ophthalmic solution, 0% dextran
  UVA Irradiation (30 mW/cm2 for 3 minutes pulsed UVA with an on/off cycle of 2 seconds UVA on/1 second UVA off)
  Laser-assisted in situ keratomileusis
- LASIK Only: Eyes assigned to this arm will receive standard LASIK with no cross-linking.
  Laser-assisted in situ keratomileusis
Period: Overall Study
Arm/Group | LASIK Followed by Cross-linking (Continuous Wave) | LASIK Followed by Cross-linking (Pulsed) | LASIK Only
Started | 0 | 2 | 0
Completed | 0 | 2 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LASIK Followed by Cross-linking (Continuous Wave) | LASIK Followed by Cross-linking (Pulsed) | LASIK Only | Total
Number analyzed (Participants) | 0 | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 |  | 0
  Between 18 and 65 years |  | 2 |  | 2
  >=65 years |  | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 |  | 1
  Male |  | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0
  Asian |  | 0 |  | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0
  Black or African American |  | 0 |  | 0
  White |  | 2 |  | 2
  More than one race |  | 0 |  | 0
  Unknown or Not Reported |  | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: MRSE Regression
Description: The co-primary efficacy endpoints are a comparison of MRSE regression in the refractive outcome between the LASIK only eyes and the LASIK with cross-linking eyes within each treatment type and duration (2 minutes continuous UVA or 3 minutes pulsed UVA cross-linking) expressed as the change between one week and six months, and one week and twelve months.
Time Frame: one week to six months
Population: This trial had extremely low enrollment due to difficulties recruiting patients therefore no analysis was conducted. Data for MSRE were collected for the two treated patients the primary endpoint is a comparison between the treatment groups. The two patients were in the same treatment group so a comparison between groups is not possible.
Arm/Group | LASIK Followed by Cross-linking (Continuous Wave) | LASIK Followed by Cross-linking (Pulsed) | LASIK Only
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: MRSE Regression
Description: as for outcome 1
Time Frame: one week to twelve months
Population: This trial had extremely low enrollment due to difficulties recruiting patients therefore no analysis was conducted.
Arm/Group | LASIK Followed by Cross-linking (Continuous Wave) | LASIK Followed by Cross-linking (Pulsed) | LASIK Only
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | LASIK Followed by Cross-linking (Continuous Wave) | LASIK Followed by Cross-linking (Pulsed) | LASIK Only
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LASIK Followed by Cross-linking (Continuous Wave) (N=0) | LASIK Followed by Cross-linking (Pulsed) (N=2) | LASIK Only (N=2)
Vision blurred (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
Foreign body sensation in eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal flap complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site has the right to publish or communicate study results upon the earlier of: (a) publication of a multi-center publication of the Study results coordinated by Sponsor; or (b) submission of the Study data by Sponsor to the FDA; provided that the Sponsor reviews the proposed communication of results within ninety (90) days in advance of its release. Sponsor can request delay of publication or data release to allow for filing of patent application prior to the publication or release.